CLINICAL TRIAL: NCT04920071
Title: Quantifying the Disease Signal to Measurement Noise Ratio With the Moorfields Acuity Chart in Age-related Macular Disease
Brief Title: Optimising Visual Acuity Measurement in Macular Degeneration
Acronym: OPTIMISE
Status: Completed | Type: Observational
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: MULP1001
Record Dates: First submitted 2021-02-09; First posted 2021-06-09 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Visual Acuity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control: 150 healthy control participants
  Interventions: Device: Visual acuity and contrast sensitivity measurement
- AMD Cohort high-contrast VA group i: Better than 0.4 logMAR
  Interventions: Device: Visual acuity and contrast sensitivity measurement
- AMD Cohort high-contrast VA group ii: 0.4-0.6 logMAR
  Interventions: Device: Visual acuity and contrast sensitivity measurement
- AMD Cohort high-contrast VA group iii: 0.6-0.8 logMAR
  Interventions: Device: Visual acuity and contrast sensitivity measurement
- AMD Cohort high-contrast VA group iv: 0.8-1.0 logMAR
  Interventions: Device: Visual acuity and contrast sensitivity measurement

INTERVENTIONS:
Device: Visual acuity and contrast sensitivity measurement — Those subjects who meet the inclusion criteria will undergo the study tests. These measurements will be performed on one eye only. Visual acuity will be quantified using two forms of the MAC chart (MAC 1 and 2) and two forms of a conventional letter design chart (C1 and 2). Contrast sensitivity will be measured using the two forms of the Pelli-Robson chart (CS1 and CS2). The order with which the test charts will be presented, in addition to the charts used (i.e. MAC 1 or 2, C1 or 2, and CS1 or 2), will be selected at random. Finally, a measurement of eye length will be collected using an IOL Master (Carl-Zeiss Meditec, USA).

SUMMARY:
Age-related macular degeneration (AMD) is the leading cause of visual impairment in the UK. The condition is characterised by damage to the region of the retina (macula) responsible for detailed central vision, this leading to problems with tasks such as reading and face-recognition. The ability to accurately measure vision is central to the detection and management of AMD. The most common test (visual acuity) typically requires patients to identify black letters of varying size on a white background, with the smallest letter read representing the limit of vision. Conventional tests are however known to be variable, making it difficult to determine if a true change in vision has occurred.

Previous work has found the Moorfields Acuity Chart, which contains specially constructed letters composed of a black core and white border, to be more sensitive to early AMD compared to standard charts. Despite this advantage, it is unclear if there is an associated increase in measurement variability with the Moorfields Acuity Chart and if this changes with the severity of disease. In this study, the relationship between vision test sensitivity and measurement variability will be quantified with both conventional visual acuity tests and the new Moorfields Acuity Chart to identify the optimal vision test to detect and monitor AMD in the clinic.

ELIGIBILITY:
Group 2 - Healthy control participants:

Inclusion criteria will include:

* Absence of ocular disease in either eye
* Male or female, aged 18 years or older
* The absence of significant media opacities
* Ability to understand nature/purpose of the study and to provide informed consent
* Ability to follow instructions and complete the study
* Ability to speak English

Exclusion criteria will include:

* Any systemic disease likely to affect visual performance
* Presence of any ocular disease
* Hearing impairment sufficient to interfere with hearing instructions
* Poor understanding of English language and/or alphabet
* Any condition which, in the investigator's opinion, would conflict or otherwise prevent the subject from complying with the required procedures, schedule, or other study conduct.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with reduced vision attributable to AMD will be recruited and tested as part of this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Ratio of disease signal (test sensitivity) to measurement noise (variability) in AMD with conventional and Moorfields Acuity Charts | 2 years
  The disease signal to measurement noise ratio (SNR) is defined as the ratio of AMD test sensitivity to the degree of measurement variability for each chart investigated in this study.

SECONDARY OUTCOMES:
Test-retest variability for the Moorfields Acuity Chart and conventional logMAR visual acuity tests | 2 years
  Measurement variability (difference in two measures captured using the same vision test on the same day) will be quantified for each vision test used in this study. This analysis will also be undertaken for participants with a range of AMD related vision loss.

CONTACTS AND LOCATIONS:
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom